CLINICAL TRIAL: NCT04965454
Title: Clinical Trial of Biomarkers for Predicting Immunotherapy Response in Hepatocellular Carcinoma
Brief Title: Evaluation of Treatment Predictors Reflecting Beta-catenin Activation in Hepatocellular Carcinoma
Acronym: ExTRACT-HCC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Queen's Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Sandi Kwee, Program Director, PET Research, Queen's Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RA-2021-018; R01CA262460 (NIH)
Record Dates: First submitted 2021-07-07; First posted 2021-07-16 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Hepatocellular Carcinoma Non-resectable
Keywords: hepatocellular carcinoma; immunotherapy; positron emission tomography; mutation profiling; liquid biopsy; personalized medicine; diagnostic; fluorocholine; immune checkpoint inhibitor
MeSH Terms: conditions — Carcinoma, Hepatocellular; Disease | interventions — fluorocholine

STUDY DESIGN:
Intervention Model Description: prospective open-label single-arm diagnostic clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Tested with Biomarkers (Experimental): For this single arm study, all enrolled subjects will undergo diagnostic testing with FCH PET/CT and genomic liquid biopsy before treatment involving an immune checkpoint inhibitor agent. A fluorine-18 fluorodeoxyglucose (FDG) PET/CT may also be performed before treatment and after 8 weeks if the pre-treatment FCH PET/CT shows low or heterogeneous tumor uptake.
  Interventions: Combination Product: Fluorine-18 fluorocholine

INTERVENTIONS:
Combination Product: Fluorine-18 fluorocholine — 18F-fluorocholine is a radiopharmaceutical imaging agent intended for use only with positron emission tomography (PET) imaging. PET with in-line computed tomography imaging of the torso will be performed following intravenous administration of a single unit dose of this investigational new drug.
  Other Names: 18F-fluorocholine; Fluorocholine; 18F-FCH; FCH; [18F]fluorocholine

SUMMARY:
This prospective clinical trial will evaluate PET/CT and genomic liquid biopsy based biomarkers as predictors of clinical therapeutic response to immune-checkpoint inhibitor (ICI) therapy for patients with inoperable hepatocellular carcinoma (HCC). The primary objective of this diagnostic trial is to assess the accuracy of pre-treatment fluorine-18 (18F-) fluorocholine (FCH) PET/CT for predicting a lack of objective response (LOR) after 16 weeks of ICI therapy.

DETAILED DESCRIPTION:
This is a prospective open-label single-arm diagnostic clinical trial evaluating fluorine-18 fluorocholine (FCH) PET/CT and cell-free DNA mutation profiling (also referred to as genomic liquid biopsy) as diagnostic tools for predicting therapeutic response in advanced HCC patients receiving immune-checkpoint inhibitor (ICI) therapy. All enrolled subjects will undergo diagnostic testing with FCH PET/CT and genomic liquid biopsy before ICI treatment. A fluorine-18 fluorodeoxyglucose (FDG) PET/CT may also be performed before treatment and after 8 weeks if the pre-treatment FCH PET/CT shows low or heterogeneous tumor uptake. The accuracy of tumor biomarkers based on PET/CT and liquid biopsy for predicting therapeutic outcome and disease progression will be determined using objective clinical endpoints based on the radiographic classification of treatment response by RECIST v1.1 applied to CT or MRI performed after 16 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older (no upper limit of age)
* Hepatocellular carcinoma diagnosis made histologically or radiographically in accordance to National Comprehensive Cancer Network guidelines (3.2019 version or higher)
* Does not qualify for surgical resection or locoregional therapy alone or has disease that has progressed after surgical resection and/or locoregional therapy
* Has measurable disease defined as at least one tumor lesion that can be accurately measured according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 on CT/MRI completed within past 6 weeks of eligibility screening
* Under the care of a licensed medical oncologist
* Life expectancy > 6 months
* Deemed eligible for treatment with an immune checkpoint inhibitor agent based on the treating medical oncologist's assessment of previous treatment failure, clinical/performance/virology status, and liver/renal/hematologic function.
* Child-Pugh score of 9 or less
* Creatinine clearance ≥ 40 mL/min, measured or calculated using the Cockcroft-Gault formula
* ALT and AST ≤7x upper limit of normal
* Total bilirubin ≤4 mg/dL
* Albumin ≥2.8 g/dL

Exclusion Criteria:

* Weight > 500 lbs (PET/CT limit)
* Pregnant or lactating female (those of child-bearing potential must be re-screened within 7 days prior to PET/CT imaging)
* Serious underlying medical condition that would impair patient's ability to tolerate the imaging procedure
* Concurrent treatment with a non-targeted therapeutic agent. Concurrent enrollment in an ICI-treatment trial and combination ICI treatment are allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-03-28 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Lack of Objective Response | 16 weeks
  Lack of Objective Response defined after 16 weeks as meeting criteria for either Stable Disease or Progressive Disease based on RECIST v1.1

SECONDARY OUTCOMES:
Objective Response | 16 weeks
  Objective Response defined after 16 weeks as meeting criteria for either Partial Response or Complete Response based on RECIST v1.1
Disease Control | 16 weeks
  Disease Control defined after 16 weeks as meeting criteria for either Partial Response, Complete Response, or Stable Disease based on RECIST v1.1

CONTACTS AND LOCATIONS:
Overall Officials: Sandi A Kwee, MD, PhD, Principal Investigator — The Queen's Medical Center
Locations (1):
- The Queen's Medical Center, Honolulu, Hawaii, United States

IPD SHARING:
Plan to Share IPD: Yes
Limited de-identified genomic and phenotypic individual participant data will be made available after the end of the trial via the NIH database of genotypes and phenotypes (dbGaP) in accordance with the NIH Genomic Data Sharing Policy. The individual level data made available by dbGaP is safeguarded by a process of controlled-access with data use limitations to be determined.
Supporting Information: ICF
Time Frame: Starting 6 months after last publication at conclusion of the trial.
Access Criteria: Controlled-Access. Contact NIH dbGaP for more information.
URL: https://www.ncbi.nlm.nih.gov/gap/

DOCUMENTS (1):
  • Informed Consent Form (2021-08-17): https://cdn.clinicaltrials.gov/large-docs/54/NCT04965454/ICF_002.pdf